CLINICAL TRIAL: NCT04386863
Title: Taxonomy of Neurorehabilitation Treatments and Outcome Measures: a Multicentre Italian Study
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: IRCCS San Camillo, Venezia, Italy (Other); Universita degli Studi di Genova (Other); AIAS di Milano Onlus (Unknown); Ospedale San Carlo Borromeo (Other); Azienda Universitaria Integrata Giuliano Isontina, Trieste, Italy (Unknown); Presidio Ospedaliero San Camillo di Torino (Unknown); Ospedali Riuniti Ancona (Other); Istituto Don Orione, Pescara, Italy (Unknown)
Responsible Party: Principal Investigator, Davide Cattaneo, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: Taxonomy
Record Dates: First submitted 2019-12-09; First posted 2020-05-13 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis; Stroke; Parkinson Disease
Keywords: Multiple Sclerosis; Stroke; Parkinson; Taxonomy; Rehabilitation; Outcome measures
MeSH Terms: conditions — Multiple Sclerosis; Stroke; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aims of the observational study are to taxonomize the contents of rehabilitation understanding goals and treatments provided to people with Parkinson Disease(PD) and Multiple Sclerosis(MS) and Stroke and their impact on the outcomes

DETAILED DESCRIPTION:
In recent years, neurological rehabilitation focused on evaluating patient's problems, with no rationalization of therapeutic interventions. Few researches investigated the contribution of the components of a neurorehabilitation program to the clinical outcome in everyday clinical practice. Moreover, there is no a standard method to categorize rehabilitative interventions, making difficult to explain why subjects improve and which of the various treatments is more effective. Thus, it was decided to build a multicentre network to collect data using a taxonomy tool developed to provide information on the goals of rehabilitation and to categorize rehabilitation interventions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Diagnosis of Parkinson Disease
* Diagnosis of Stroke
* Participants' rehabilitation program must include at least 10 sessions of physical therapy.

Exclusion Criteria:

- Unable to understand the aim of the study or unable to sign the informed consent form;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in all the centers involved in the study, including both inpatients and outpatients.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Change in Two minute walking test | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  The Two minute walking test is a test used to evaluate functional exercise capacity. Subjects are instructed to walk as fast as possible in 2 minutes, along a 30-m hallway. Total distance walked is recorded
Change in Box and Blocks test | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  The Box and Block Test measures unilateral gross manual dexterity. The test consists of a box with a partition in the middle and is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial.

SECONDARY OUTCOMES:
Change in Reaching Performance Scale | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  The Reaching Performance Scale is a visual scale used in clinics to provide assessment of motor capabilities during reaching movements. It was designed to investigate reaching movements at low height in the workspace of the limb, at increasing distance. Higher scores indicate better performances.
Change in Activities-specific Balance Confidence scale | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  The Activities-specific Balance Confidence scale asks individuals to self-report their balance confidence in successfully performing 16 specific movement activities of varied balance difficulty. Higher scores indicate better balance confidence.
Change in Cognitive dual-task Timed-Up-and-Go test | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  Patients will be first asked to stand from a seated position, walk 3 m at their usual pace, turn around, walk back to the chair, and sit down (the Timed Up and Go test). Walking aids were allowed. After a recovery phase, patients will be asked to perform the same exercise while performing a cognitive dual task (continuously subtracting 2, starting from 100; the Cognitive dual-task Timed Up and Go test). Lower times indicate better performances.
Change in Manual Ability Measurement | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  The Manual Ability Measurement is a questionnaire on perceived ease or difficulty that a persons may experience when performing unilateral and bilateral ADL tasks. Higher scores indicate less difficulty in ADL tasks.
Change in modified Dynamic Gait Index | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  The modified Dynamic Gait Index is a clinical outcome measure to assess the ability to modify and adapt gait and balance during complex walking tasks. Higher scores indicate better performances.
Modified Barthel Index | Baseline and after a minimum of 2 weeks up to a maximum of 20 weeks
  Measure of physical disability used widely to assess behaviour relating to activities of daily living for patients with disabling conditions. It measures what patients do in practice. Higher scores indicate low level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattaneo, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (7):
- Italy (7):
  - Universita degli Studi di Genova, Genova
  - Fondazione Don Gnocchi ONLUS, Milan
  - Ospedale San Carlo Borromeo, Milan
  - AIAS di Milano Onlus, Milan
  - Ospedale San Giovanni Battista ACISMOM, Roma
  - Università degli studi di Trieste, Trieste
  - IRCCS San Camillo, Venice

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dijkers MP, Hart T, Tsaousides T, Whyte J, Zanca JM. Treatment taxonomy for rehabilitation: past, present, and prospects. Arch Phys Med Rehabil. 2014 Jan;95(1 Suppl):S6-16. doi: 10.1016/j.apmr.2013.03.032. PMID 24370326
- [Background] Rasova K, Freeman J, Martinkova P, Pavlikova M, Cattaneo D, Jonsdottir J, Henze T, Baert I, Van Asch P, Santoyo C, Smedal T, Beiske AG, Stachowiak M, Kovalewski M, Nedeljkovic U, Bakalidou D, Guerreiro JM, Nilsagard Y, Dimitrova EN, Habek M, Armutlu K, Donze C, Ross E, Ilie AM, Martic A, Romberg A, Feys P. The organisation of physiotherapy for people with multiple sclerosis across Europe: a multicentre questionnaire survey. BMC Health Serv Res. 2016 Oct 6;16(1):552. doi: 10.1186/s12913-016-1750-6. PMID 27716390
- [Background] Dejong G, Horn SD, Gassaway JA, Slavin MD, Dijkers MP. Toward a taxonomy of rehabilitation interventions: Using an inductive approach to examine the "black box" of rehabilitation. Arch Phys Med Rehabil. 2004 Apr;85(4):678-86. doi: 10.1016/j.apmr.2003.06.033. PMID 15083447